CLINICAL TRIAL: NCT06139965
Title: Validity and Reliability of the Turkish Version of the Comprehensive Coordination Scale in Parkinson's Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Gokce Yagmur Gunes Gencer, Assist.Prof, Akdeniz University
Other Study IDs: KAEK-633
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Comprehensive Coordination Scale; Validity; Reliability
MeSH Terms: conditions — Parkinson Disease | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validity and Reliability — Assessment study

SUMMARY:
The aim of this study is to investigate the Turkish adaptation of the Comprehensive Coordination Scale and its validity and reliability in Parkinson's patients.

DETAILED DESCRIPTION:
A Turkish version of the Comprehensive Coordination Scale will be made. Then, Comprehensive Coordination Scale, 9-Hole Peg Test, Timed Up and Go Test, Berg Balance Scale, Functional Reaching Test and Modified Hoehn and Yahr Scale will be applied to patients with Parkinson's, respectively. In order to determine the reliability of the scale, only the "Comprehensive Coordination Scale" will be video recorded during the first evaluation and inter-rater reliability will be performed by another physiotherapist. For test-retest reliability, patients will be evaluated seven days later by the first physiotherapist who made the evaluation by watching the video again.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's,
* Mini mental test score over 24,
* Those who have not experienced any serious neurological or orthopedic problems in the last 6 months,
* İndividuals who agreed to participate in the study

Exclusion Criteria:

* Mini mental test score <24,

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-01-05 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Coordination Scale | Baseline (First assessment)
  The Comprehensive Coordination Scale (CCS) is a measure of coordination of multiple body segments at both motor performance (endpoint movement) and quality of movement (joint rotations and interjoint coordination) levels based on observational kinematics.

SECONDARY OUTCOMES:
9 Hole Peg Test | Baseline (First assessment)
  The Nine-Hole Peg Test (9-HPT) is a standardized, quantitative assessment used to measure finger dexterity.
Timed Up and Go Test (TUG) | Baseline (First assessment)
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults.
Berg Balance Test | Baseline (First assessment)
  The Berg Balance Scale (BBS) is a 14-item objective measure that assesses static balance and fall risk in adults.
Functional Reach Test | Baseline (First assessment)
  The Functional Reach Test assesses a patient's stability by measuring the maximum distance an individual can reach forward while standing in a fixed position.
Modified Hoehn and Yahr Scale | Baseline (First assessment)
  The Hoehn and Yahr scale is used to describe the symptom progression of Parkinson disease

CONTACTS AND LOCATIONS:
Overall Officials: Gökçe Yağmur Güneş Gencer, Assist.Prof., Principal Investigator — Akdeniz University; Lütfiye Akkurt, Assist.Prof., Study Chair — Kutahya Health Sciences University; Hayri Aktaş, MSc, Study Chair — Akdeniz University; Nazan Ş Erdem, MD, Study Chair — Özel Termessos Hastanesi
Locations (2):
- Turkey (Türkiye) (2):
  - Gokce Yagmur Gunes Gencer, Antalya
  - Ozel Termessos Hastanesi, Antalya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alouche SR, Molad R, Demers M, Levin MF. Development of a Comprehensive Outcome Measure for Motor Coordination; Step 1: Three-Phase Content Validity Process. Neurorehabil Neural Repair. 2021 Feb;35(2):185-193. doi: 10.1177/1545968320981955. Epub 2020 Dec 22. PMID 33349134